CLINICAL TRIAL: NCT00259662
Title: High-dose Statin Therapy in the Perioperative Period and DVT Prevention.
Brief Title: High-dose Periop Statins for Prevention of DVT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Washington Mutual Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: HIC0507000393
Record Dates: First submitted 2005-11-28; First posted 2005-11-29 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Gynecologic Oncological Pelvic/Abdominal Surgery
Keywords: cancer--ovarian; cancer--endometria; deep vein thrombosis; statin therapy in perioperative period
MeSH Terms: conditions — Ovarian Neoplasms; Venous Thrombosis | interventions — Atorvastatin

INTERVENTIONS:
Drug: atorvastatin

SUMMARY:
This study is designed to determine if the use of atorvastatin (Lipitor), a member of the HMG coA reductase inhibitor class of drugs referred to as statins, will reduce inflammatory responses and deep vein thrombosis formation when given in high doses in the perioperative period.

ELIGIBILITY:
Inclusion Criteria:

* gynecologic tumor scheduled for resection

Exclusion Criteria:

* prior reaction to statins
* renal insufficiency
* liver disease
* h/o alcoholism
* prior h/o DVT or hypercoagulability
* concurrent medications that significantly affect cytochrome P450 3A4
* breast feeding or pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2005-11; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Decrease in incidence of deep vein thrombosis

SECONDARY OUTCOMES:
Decrease in inflammatory mediator release.

CONTACTS AND LOCATIONS:
Overall Officials: Ala S Haddadin, MD, Principal Investigator — Assistant Professor
Locations (1):
- Yale-New Haven Hospital, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Lippi G, Favaloro EJ, Sanchis-Gomar F. Venous thrombosis associated with HMG-CoA reductase inhibitors. Semin Thromb Hemost. 2013 Jul;39(5):515-32. doi: 10.1055/s-0033-1343892. Epub 2013 Apr 29. PMID 23629822